CLINICAL TRIAL: NCT01872104
Title: Longterm Outcome of Photodynamic Therapy Compared With Chemotherapy Alone in Patients With Advanced Rectal Cancer
Brief Title: Safety and Efficiency of Photodynamic Therapy for Rectal Cancer
Acronym: PDT-R-01
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Modifying the clinnicaltrials
Sponsor: li xiong (Other)
Responsible Party: Sponsor-Investigator, li xiong, Doctor, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDT-R-01; PDT-R-01 (Other: Central South University)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Rectal Cancer
Keywords: rectal cancer; rectal adenocarcinoma; photodynamic therapy; chemothrapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy alone (No Intervention): Group that be scheduled to undergo chemothrapy only using FOLFOX4 protocol.
- PDT and Chemotherapy (Experimental): Group that not only be scheduled to undergo chemothrapy using FOLFOX4 protocol,but also receive colonscopy-assisted PDT.
  Interventions: Procedure: Photodynamic therapy

INTERVENTIONS:
Procedure: Photodynamic therapy — Each patient to whom PDT was offered underwent a specific, detailed educational process by a dedicated team member(P.B., P.J., or K.E.), after which informed consent was obtained.Porfimer sodium (Photofrin; Axcan Pharma Inc, Quebec, Canada)was used as a photo sensitizing agent, administered intravenously at a dose of 2 mg/kg body weight 48 hours before illumination.A diode laser system (InGaAIP Laser Diode; Diomed Inc, An-dover, MA) with a maximum power output of 2000 mW and a wavelength of 633+-3 nm was used as a light source, delivered through a 3.0-m length fiber having a 2.5-cm-long cylindrical diffuser at its distal end (Pioneer Optics, Windsor Locks, CT).
  Arms: PDT and Chemotherapy

SUMMARY:
This research is a prospective randomized controlled trial.It aimed to determine longterm outcomes and factors associated with increased survival after photodynamic therapy (PDT) through colonscopy compared with chemotherapy alone in patients presenting with advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with advanced rectal cancer 2.Patients are willing to join in this clinical trial.

Exclusion Criteria:

* 1.Patients with advanced rectal cancer can not suffer PDT procedure. 2.Allergy to photosensitizer

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Survival rate | one month

SECONDARY OUTCOMES:
Progression-free survival | One month

OTHER OUTCOMES:
Quality of life | one month

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Result] Allison RR, Sheng C, Cuenca R, Bagnato VS, Austerlitz C, Sibata CH. Photodynamic therapy for anal cancer. Photodiagnosis Photodyn Ther. 2010 Jun;7(2):115-9. doi: 10.1016/j.pdpdt.2010.04.002. Epub 2010 May 7. PMID 20510306